CLINICAL TRIAL: NCT05138458
Title: A Phase 1/2, Open-Label, First-in-human, Multiple Ascending Dose Multicenter Study of MT-101 in Subjects With CD5+ Relapsed/Refractory T Cell Lymphoma
Brief Title: A Study of MT-101 in Subjects With CD5+ Relapsed/Refractory TCL
Acronym: IMAGINE
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Temporary operational pause; no safety concerns.
Sponsor: Myeloid Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MTX-TCL-101
Record Dates: First submitted 2021-11-16; First posted 2021-12-01 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Lymphoma, T-Cell, Peripheral; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Adoptive Cellular Immunotherapy; Cell Therapy
Keywords: T Cell Lymphoma; PTCL; CTCL; MF; MT-101; CD5 chimeric antigen receptor; Myeloid cells; Monocytes; Chimeric Antigen Receptor; CAR Monocyte Therapy
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Lymphoma, T-Cell | interventions — Drug Therapy

STUDY DESIGN:
Intervention Model Description: Multi-ascending dose escalation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 and Cohort 3 (Experimental): MT-101
  Interventions: Biological: MT-101
- Cohort 2 and Cohort 4 (Experimental): MT-101 preceded by conditioning (lymphodepleting) chemotherapy
  Interventions: Other: MT-101 + Conditioning (Lymphodepleting) Chemotherapy

INTERVENTIONS:
Biological: MT-101 — CD5 ATAK cells
  Arms: Cohort 1 and Cohort 3
Other: MT-101 + Conditioning (Lymphodepleting) Chemotherapy — IV administration of fludarabine and cyclophosphamide
  Arms: Cohort 2 and Cohort 4

SUMMARY:
This is a Phase 1/2 study to test the safety, tolerability, and efficacy of the investigational agent MT-101 in patients with T cell Lymphoma. MT-101 is made with myeloid cells collected from the patient's blood. The myeloid cells are modified and later infused back into their veins. The modified myeloid cells recognize the tumor cells and are designed to target and kill them.

DETAILED DESCRIPTION:
The research study is divided into two parts. The first part will be to determine the safety and tolerability of the study drug product. During this part of the study, there will be 4 groups of study patients. The first group of patients will receive a low dose of cells, the second group will receive the low dose of cells and lymphodepleting chemotherapy to reduce the number of T cells in the blood, the third group will receive a higher dose of cells, and the fourth group will receive the higher dose of cells and lymphodepleting chemotherapy to reduce the number of T cells in the blood. In the second part of the study, cells with or without chemotherapy will be administered based on results of Part 1 and the safety, tolerability, and efficacy of MT-101 will be assessed. All patient groups will receive 6 doses of drug product over 3 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

* Adults age > or equal to18 at the time the Informed Consent is signed
* Refractory or relapsed pathologically confirmed T Cell Lymphoma (TCL): Peripheral T cell Lymphoma not otherwise specified (PTCL-NOS) , Angioimmunoblastic T cell Lymphoma (AITL), ALK-negative anaplastic large cell lymphoma (ALCL), ALK-positive ALCL, or Mycosis Fungoides (MF) stage IIB-IV including large cell transformation
* CD5-expressing tumor by IHC or flow cytometry of tumor biopsy within 3 months of Screening or at Screening
* Eastern Cooperative Oncology Group performance status < 2
* Adequate organ function as defined in the protocol.

Key Exclusion Criteria:

* B1 and B2 disease (as defined in protocol for subjects with MF)
* Known central nervous system involvement by PTCL
* History of allogeneic transplant
* History of intolerance to leukapheresis, plasmapheresis, or blood donation
* Pregnant or nursing women
* Any acute illness including fever (> 100.4°F or > 38°C), except fever related to tumor
* Active systemic bacterial, fungal, or viral infection
* Active chronic infection
* Other primary malignancies, except adequately treated malignancies or complete remission
* Active autoimmune disease that has required systemic therapy in the last 2 years
* History of hemophagocytic lymphohistiocytosis
* History of severe, immediate hypersensitivity reaction attributed to penicillin
* Any other condition that, in the opinion of the Investigator, would make the subject unsuitable for the study or unable to comply with the study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability of MT-101 | 4 weeks
  Safety and tolerability of the drug will be determined based on observed adverse events (AEs), including all potential dose limiting toxicities.

SECONDARY OUTCOMES:
MT-101 cell kinetics in blood | 4 weeks
  The quantity of MT-101 RNA in the blood.
The objective response rate | 24 weeks
  The ORR is defined as the number (%) of subjects achieving a best overall response of complete response (CR) or partial response (PR)

OTHER OUTCOMES:
Duration of response (DOR) | 48 weeks
  DOR is the time interval between the date of first assessment of PR or CR to the date of the follow-on first documentation of progressive disease or death, whichever occurs earlier.
Progression free survival (PFS) | 48 weeks
  PFS is defined as the time from the date of the first administration of MT-101 to the date of first documentation of progressive disease or death, whichever occurs earlier.
Overall survival (OS) | 48 weeks
  OS is defined as the time from date of the first administration of MT-101 to the date of death.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Gerber, MD, MPH, Study Director — Myeloid Therapeutics
Locations (6):
- United States (6):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Dana-Farber/Mass General Brigham Cancer Care, Boston, Massachusetts
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Virginia Comprehensive Cancer Center, Charlottesville, Virginia